CLINICAL TRIAL: NCT00917774
Title: A Gender-Specific Posterior Cruciate-Substituting High-Flexion Knee Prosthesis Does Not Improve Fit and Function Compared With a Standard Posterior Cruciate-Substituting High-Flexion Knee Prostheis A Prospective, Randomized Study
Brief Title: A Gender-Specific Posterior Cruciate-Substituting High-Flexion Knee Prosthesis Does Not Improve Fit and Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Young-Hoo, Kim M.D., Ewha Womans University Mokdong Hospital Joint Replacement Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-6-10
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Osteoarthritis of the Knee; Female
Keywords: gender specific knee; osteoarthritis; total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard LPS Flex (Active Comparator): Nexgen LPS-Flex total knee design used for TKA
  Interventions: Device: Standard LPS flex TKA
- Gender specific LPS-Flex (Experimental): Gender specific LPS flex design used for TKA in female patients
  Interventions: Device: Gender specific LPS -Flex TKA

INTERVENTIONS:
Device: Standard LPS flex TKA — TKA by Standard LPS flex TKA
  Other Names: Standard Zimmer Nexgen Legacy posterior stabilized High-flex
  Arms: Standard LPS Flex
Device: Gender specific LPS -Flex TKA — Total knee design created specific for female patients
  Other Names: Gender specific Zimmer LPS High-flex
  Arms: Gender specific LPS-Flex

SUMMARY:
The purpose of this study was to compare functional and radiographic results, range of motion of the knee, patient satisfaction, femoral component, revision and complication rates in patients receiving either a standard posterior cruciate substituting-flex (LPS-flex) or gender-specific posterior cruciate substituting-flex (LPS-Flex) total knee prosthesis.

DETAILED DESCRIPTION:
Recently much debate and discussion has focused on the effect of gender-specific total knee arthroplasty. The purpose of this study was to compare functional and radiographic results, range of motion of the knee, patient satisfaction, femoral component, revision and complication rates in patients receiving either a standard posterior cruciate substituting-flex (LPS-flex) or gender-specific posterior cruciate substituting-flex (LPS-Flex) total knee prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* End-stage osteoarthritis of the knee joint requiring total knee arthroplasty with bilateral disease, in female patients

Exclusion Criteria:

* Male patient
* Inflammatory disease
* patient with other Lower extremity disease which may affect functional outcome
* Neurologic disease effecting patients lower extremity
* Revision surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2006-11; Primary Completion 2007-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
knee function | 2 years

SECONDARY OUTCOMES:
implant fit to patient | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Yoowang Choi, MD, Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea